CLINICAL TRIAL: NCT06188702
Title: A Phase 1/2, Open-label, Multicenter Clinical Trial Investigating the Safety, Tolerability, Pharmacokinetics, and Antineoplastic Activity of S095035 (MAT2A Inhibitor) as a Single Agent and in Combination in Adult Participants With Advanced or Metastatic Solid Tumors With Homozygous Deletion of MTAP
Brief Title: S095035 as a Single Agent and in Combination in Adult Participants With Advanced or Metastatic Solid Tumors With Deletion of MTAP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Servier Bio-Innovation LLC (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other); Tango Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95035-001; 2025-521249-25-00 (EU CTIS Number)
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: MTAP-deleted Solid Tumors
Keywords: MAT2A; MTAP; Solid Tumors; PRMT5; SAM; Synthetic Lethality; MTAP deletion; MAT2A Inhibitor; Advanced Solid Tumors; Biliary Tract Cancer; Non-small Cell Lung Cancer; Pancreatic Adenocarcinoma; Gastroesophageal Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase 1 Arm 1 - S095035 single-agent dose escalation (Experimental)
  Interventions: Drug: S095035
- Phase 1 Arm 2 - S095035-TNG462 combination dose escalation (Experimental)
  Interventions: Drug: S095035; Drug: TNG462
- Phase 2 Arm 1a NSCLC - S095035 single-agent dose expansion (Experimental): Non-Small Cell Lung Cancer
  Interventions: Drug: S095035
- Phase 2 Arm 1b BTC - S095035 single-agent dose expansion (Experimental): Biliary Tract Cancer
  Interventions: Drug: S095035
- Phase 2 Arm 1c PDAC - S095035 single-agent dose expansion (Experimental): Pancreatic Ductal Adenocarcinoma
  Interventions: Drug: S095035
- Phase 2 Arm 1d Basket arm - S095035 single-agent dose expansion (Experimental)
  Interventions: Drug: S095035
- Phase 2 Arm 2a BTC - S095035-TNG462 combination dose expansion (Experimental): Biliary Tract Cancer
  Interventions: Drug: S095035; Drug: TNG462
- Phase 2 Arm 2b Gastroesophageal - S095035-TNG462 combination dose expansion (Experimental)
  Interventions: Drug: S095035; Drug: TNG462
- Phase 2 Arm 2c PDAC - S095035-TNG462 combination dose expansion (Experimental): Pancreatic Ductal Adenocarcinoma
  Interventions: Drug: S095035; Drug: TNG462

INTERVENTIONS:
Drug: S095035 — S095035 will be taken orally every day in 28-day cycles.
Drug: TNG462 — TNG462 will be taken orally every day in 28-day cycles.
  Arms: Phase 1 Arm 2 - S095035-TNG462 combination dose escalation; Phase 2 Arm 2a BTC - S095035-TNG462 combination dose expansion; Phase 2 Arm 2b Gastroesophageal - S095035-TNG462 combination dose expansion; Phase 2 Arm 2c PDAC - S095035-TNG462 combination dose expansion

SUMMARY:
This is a first-in-human Phase 1/2, multicenter, open-label study of S095035 as single-agent, or in combination with TNG462 in adult participants with advanced or metastatic solid tumors with homozygous deletion of MTAP who have failed to respond to or have progressed after at least 1 prior treatment regimen, and for whom additional effective standard treatment is not available. S095035 is an oral methionine adenosyltransferase 2A [MAT2A] inhibitor. TNG462 is a protein arginine N-methyltransferase 5 [PRMT5] inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Estimated life expectancy ≥3 months.
* ECOG PS 0-1
* Participants able to comply with highly effective method of birth control requirements.
* Participants with histologically confirmed advanced or metastatic solid tumor's (excluding central nervous system tumors other than IDHwt glioblastoma), with measurable disease as per RECIST 1.1 or RANO 2.0 criteria for participants with IDHwt glioblastoma, that have progressed after at least one prior treatment regimen given for advanced/metastatic disease, and for whom additional effective standard therapy is not available. Patients in China with IDHwt glioblastoma will not be included.
* Participants with pre-existing documented MTAP homozygous gene deletion in their tumor tissue, determined using a next generation sequencing in vitro diagnostic test prior to screening.
* Phase 1 only - Participants (except IDHwt glioblastoma) willing to undergo paired fresh biopsy (pre-treatment and on-treatment) procedure. Exceptions may be made for feasibility and safety concerns. IDHwt glioblastoma must provide archival tissue from most recent surgery or biopsy.
* Adequate organ functions.
* Phase 2 only - Participants in dose expansion, except those with IDHwt glioblastoma, must provide newly collected tumor biopsies at screening. If not medically feasible archival tissue may be used, provided it was collected within 3 months before study entry and no treatment has been received since the most recent biopsy.
* Phase 2 only - Participants with IDHwt glioblastoma must provide archival tissue from their most recent surgery or biopsy, collected before screening.
* Phase 2 only - Participants in China who are to be considered for enrollment in the single agent dose expansion Arms and who have a pre-existing, documented cyclin-dependent kinase inhibitor 2A (CDKN2A) homozygous gene deletion in their tumor tissue (confirmed by an NGS IVD test), but do not have homozygous MTAP deletion reported, will need to be pre-screened to confirm homozygous MTAP deletion. Pre screening for homozygous MTAP deletion will be conducted using a central NGS IVD test using an archival tumor tissue, preferably the most recent and not older than 3 years.
* Phase 2 Arm 1a only - Participants with histologically or cytologically confirmed metastatic or unresectable locally advanced NSCLC with homozygous deletion of MTAP, with measurable disease as per RECIST version 1.1, who have progressed or experienced disease recurrence during or after at least 1 prior line of standard-of-care systemic therapy in the advanced/metastatic setting.
* Phase 2 Arm 1b only - Participants with histologically or cytologically confirmed metastatic or unresectable locally advanced BTC with homozygous deletion of MTAP, who have progressed or experienced disease recurrence during or after at least 1 prior line of standard-of-care systemic therapy in the advanced/metastatic setting.
* Phase 2 Arm 1c only - Participants with histologically or cytologically confirmed metastatic or unresectable locally advanced PDAC with homozygous deletion of MTAP, who have progressed or experienced disease recurrence during or after at least 1 prior line of standard-of-care systemic therapy in the advanced/metastatic setting.
* Phase 2 Arm 1d only - Participants with any other locally advanced or metastatic malignancies with homozygous deletion of MTAP, who have received and progressed of experienced recurrence during or after receiving at least 1 prior line of standard-of-care systemic therapy in the advanced/metastatic setting.
* Phase 2 Arm 2a only - Participants with histologically or cytologically confirmed metastatic or unresectable locally advanced BTC with homozygous deletion of MTAP, who have progressed or experienced disease recurrence during or after receiving at least 1 prior line of standard-of care systemic therapy in the advanced/metastatic setting.
* Phase 2 Arm 2b only - Participants with histologically or cytologically confirmed metastatic or unresectable locally advanced gastroesophageal cancer with homozygous deletion of MTAP, who have progressed or experienced disease recurrence during or after receiving at least 1 prior line of standard-of-care systemic therapy in the advanced/metastatic setting.
* Phase 2 Arm 2c only - Participants with histologically or cytologically confirmed metastatic or unresectable locally advanced PDAC with homozygous deletion of MTAP, who have progressed or experienced disease recurrence during or after receiving at least 1 prior line of standard-of-care systemic therapy in the advanced/metastatic setting.

Exclusion Criteria:

* Inability to take an orally administered drug, or medical disorder or prior surgical resection that may affect the absorption of the study drug.
* Active second primary malignancy other than non-melanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's Medical monitor and investigator agree and document that it should not be exclusionary.
* Known prior severe hypersensitivity to any component of the study drug formulation.
* Major surgery within 4 weeks prior to the first study drug administration or participants who have not recovered from side effects of the surgery.
* Have a known history of Gilbert's syndrome.
* Participants with a known clinically significant cardiovascular disease or condition.
* Participants with thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 4 weeks prior to first IMP administration.
* Active brain metastases.
* Participants who have received systemic anticancer treatment or radiotherapy less than 2 weeks before the first dose of study drug
* Pregnant or lactating women.
* Women of childbearing potential who have a positive pregnancy test within 7 days prior to the first day of study drug administration.
* History of gastrointestinal perforation and /or fistula or aorto-esophageal fistula within 6 months prior to first study drug intake.
* Severe or uncontrolled active acute or chronic infection.
* Participants who have already received a MAT2A or PRMT5 inhibitor.
* A medical condition that results in increased clinically significant photosensitivity (e.g., solar urticaria, lupus erythematosus, etc.).
* Participants who are scheduled to receive the S095035-TNG462 combination, with a known clinically significant ophthalmologic disease, including:
* Prior history of drug-induced or toxic retinopathy or optic neuropathy
* Uncontrolled glaucoma
* Pre-existing macular degeneration
* Ongoing Grade ≥2 retinopathy, optic neuropathy, or optic neuritis
* Other known active retinal pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2031-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | Through cycle 1 (each cycle is 28 days)
  Phase 1 only
Total number of adverse events (AEs) | Through the Safety Follow-up Visit (until 30 days after the last dose of study treatment) approximately 5 years
  Phase 1 only
Total number of serious adverse events (SAEs) | Through the Safety Follow-up Visit (until 30 days after the last dose of study treatment) approximately 5 years
  Phase 1 only
Objective response rate (ORR) | Through the end of the study (approximately 5 years)
  Phase 2 only; Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 criteria as per the investigator's assessment and by blinded independent central review (BICR)

SECONDARY OUTCOMES:
Area under the concentration-vs-time curve (AUC) from 0 to time of last measurable concentration (AUC0-t) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
AUC from 0 to infinity (AUC0-∞) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
AUC over 1 dosing interval at steady state (AUCtau,ss) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
Time to maximum concentration (Tmax) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
Maximum concentration (Cmax) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
Trough concentration (Ctrough) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
Half-life (t½) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
Apparent volume of distribution (Vd/F) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
Apparent clearance (CL/F) | Through the last dose of study treatment (approximately 5 years)
  Phase 1 and 2
Change from baseline in plasma concentrations of S-adenosylmethionine (SAM) and/or tumor symmetric dimethylarginine (SDMA) residues during treatment | Through the last dose of study treatment (approximately 5 years)
  Phase 1 only
Objective response rate (ORR) | Through the end of the study (approximately 5 years)
  Phase 1 only; Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 criteria as per the investigator's assessment
Best overall response (BOR) | Through the end of the study (approximately 5 years)
  Phase 1 and 2; Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 criteria as per the investigator's assessment for Phase 1 and 2, and by BICR only for Phase 2.
Clinical benefit rate (CBR) | Through the end of the study (approximately 5 years)
  Phase 1 and 2; CBR=complete response [CR]+partial response [PR]+stable disease [SD] ) ≥6 months, Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 criteria as per the investigator's assessment for Phase 1 and 2, and by BICR only for Phase 2
Duration of response (DOR) | Through the end of the study (approximately 5 years)
  Phase 1 and 2; Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 criteria as per the investigator's assessment for Phase 1 and 2, and by BICR only for Phase 2. The time from date of first documented confirmed CR or confirmed PR to date of first documented disease progression or death due to any cause.
Time to response (TTR) | Through the end of the study (approximately 5 years)
  Phase 1 and 2; Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 criteria as per the investigator's assessment for Phase 1 and 2, and by BICR only for Phase 2. The time from the date of randomization to date of first documented confirmed complete response (CR) or confirmed partial response (PR).
Progression-free Survival (PFS) | Through the end of the study (approximately 5 years)
  Phase 2 Only; Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 criteria as assessed by investigator and by BICR
Overall Survival (OS) | Through the end of the study (approximately 5 years)
  Phase 2 Only; Per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 criteria as assessed by investigator and by BICR
Total number of adverse events (AEs) | Through the Safety Follow-up Visit (until 30 days after the last dose of study treatment) approximately 5 years
  Phase 2 Only
Total number of serious adverse events (SAEs) | Through the Safety Follow-up Visit (until 30 days after the last dose of study treatment) approximately 5 years
  Phase 2 Only
Number of dose interruptions | Through the last dose of study treatment (approximately 5 years)
  Phase 2 Only
Number of dose reductions | Through the last dose of study treatment (approximately 5 years)
  Phase 2 Only
Dose intensity | Through the last dose of study treatment (approximately 5 years)
  Phase 2 Only

CONTACTS AND LOCATIONS:
Locations (33):
- United States (9):
  - University of California Los Angeles, Los Angeles, California
  - University of California, San Francisco (Ucsf) School of Medicine, San Francisco, California
  - Lake Mary Cancer Center - Florida Cancer Specialists & Research Institute, Lake Mary, Florida
  - Community Health Network, Indianapolis, Indiana
  - Dana Farber Cancer Institue, Boston, Massachusetts
  - Duke University School of Medicine, Durham, North Carolina
  - Taylor Cancer Research Center, Maumee, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - NEXT Oncology, Austin, Texas
- Australia (4):
  - Scientia Clinical Research, Randwick, New South Wales
  - The Alfred, Prahran, Victoria
  - Townsville University Hospital, Douglas
  - Royal Hobart Hospital, Hobart
- Denmark (2):
  - University Hospital Rigshospitalet, Copenhagen
  - Odense Universitets Hospital, Odense
- France (2):
  - Institut Bergonié, Bordeaux
  - Centre Georges-François Leclerc, Dijon
- Germany (4):
  - Charite Universitatsmedizin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Med Fakultaet Heidelberg, Heidelberg
  - Universitätsklinikum Ulm, Ulm
- Italy (5):
  - Istituto Europeo Di Oncologia, Milan
  - A.O.U. Seconda Università Degli Studi Di Napoli, Napoli
  - Ist. Nazionale Tumori Irccs Fondazione G Pascale, Napoli
  - Instituto Clinico Humanitas Irccs, Rozzano
  - Policlinico G.B. Rossi A.O.U.I. Di Verona, Verona
- Japan (3):
  - Aichi Cancer Center, Aichi
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - The Cancer Institute Hospital of JFCR, Tokyo
- Spain (4):
  - Next Oncology-Hospital Quironsalud Barcelona, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Start Madrid Group - Hm Ciocc, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/